CLINICAL TRIAL: NCT04336813
Title: Phone-based Audience Response System as an Adjunct in Orthodontic Teaching of Undergraduate Dental Students: a Cross-over Randomised Controlled Trial
Brief Title: Phone-based Audience Response System as an Adjunct in Orthodontic Teaching of Undergraduate Dental Students
Acronym: PBAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Principal Investigator, Fahad AlHarbi, Assistant Professor, Prince Sattam Bin Abdulaziz University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 1439-03-001
Record Dates: First submitted 2020-04-03; First posted 2020-04-07 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Academic Performance
Keywords: ARS,; Audience response system; Education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Receive ARS in lecture 1 and act as controller in lecture 2
  Interventions: Other: Audience Response system
- Group b (Active Comparator): Receive ARS in lecture 2 and act as controller in lecture 1
  Interventions: Other: Audience Response system

INTERVENTIONS:
Other: Audience Response system — In the lecture hall, G1 was separated from G2, and both groups completed an assessment of written multiple-choice questions (MCQs) scored out of 20, before the lecture. During L1, phone based (ARS) questions (PB-ARS) secretly displayed on the smart phones of the students in G1, and they were allowed to read the question and answer it, while those in parallel arm of the trial (G2) were blinded to those questions and answers. At the end of L1, both groups completed the same written MCQs assessment
  Other Names: Polleverywhere

SUMMARY:
Methodology :A cross-over randomised controlled trial comparing two teaching methods Duration :Start date 6th December 2017 to 29st May 2018 Objective : To evaluate the effectiveness phone-based audience response system (PB-ARS) on knowledge retention and performance in teaching orthodontics for dental undergraduate students in a Saudi Dental School Number:The cohort of the trial includes 34 fourth-year dental students that represents whole fourth-year undergraduate class Main Inclusion criteria : whole fourth-year undergraduate class in a Saudi Dental college.

Statistical Analysis : The normal distribution will be tested. The Mann-Whitney U test will used to compare the median score for each answer that would be given by students in the questionnaires. Scores will be analyzed and compared to assess knowledge retention using cross-over analysis with Mann-Whitney U test

DETAILED DESCRIPTION:
Design:

The trial was designed as a cross-over clustered randomized control trial (each group was a cluster), so that each group acted as their own control for their knowledge's retention and perception.

Setting and consent: College of Dentistry, Prince Sattam Bin Abdulaziz University/Alkharj/ Saudi Arabia. Written consents were obtained from students before commencing the trail.

Participants : The cohort of the trial included the whole fourth-year undergraduate class (34 undergraduate dental students) in order to eliminate selection bias. Participants in this study had no prior orthodontic teaching, hence, no bias associated with increased knowledge in any orthodontic field was anticipated.

Randomization: Students were allocated to one of two even groups (G1 or G2) using computer generated randomization. each group (G1 and G2) consisted of 17 male students with a mean age of (23.27 years ± 0.86).

Intervention :

Lectures : Simultaneously, G1 and G2 attended two lectures (L1&L2): L1 was titled "Management of Class III malocclusion", L2 was titled "Management of open bite and cross-bite". Both lectures were presented at the main campus of Prince Sattam Bin Abdulaziz College of Dentistry and they were conducted in an identical manner in all aspects including:

* Presentation in PowerPoint (Microsoft Corp, Redmond, WA)
* Both lectures were delivered by the same registered specialist orthodontist (FA),
* Learning outcomes of the delivered lectures (T1 and T2) were based on teaching outcomes specified by the National Commission for Academic Accreditation and Assessment in Saudi Arabia, and
* Both lectures delivered over the same period of time. Prior to lectures, students were instructed to register with the audience response system (ARS) and download its application (Poll Everywhere, San Francisco, California, USA, https://www.polleverywhere.com). Additional smart phones were available to students who do not have smart phones at the time of the lecture. Students were unaware of their allocation until the beginning of the first lecture.

In the lecture hall, G1 was separated from G2, and both groups completed an assessment of written multiple-choice questions (MCQs) scored out of 20, before the lecture. During L1, phone based (ARS) questions (PB-ARS) secretly displayed on the smart phones of the students in G1, and they were allowed to read the question and answer it, while those in parallel arm of the trial (G2) were blinded to those questions and answers. At the end of L1, both groups completed the same written MCQs assessment . A similar protocol was undertaken during L2 a week later, except that the groups were crossed-over, hence, the group which has had ARS integrated lecture in the previous week, has received in a non-ARS integrated lecture, and vice versa.

Formative exam:

MCQs formative tests consisted of 20 questions related to the taught topics during L1 and L2 was undertaken. In order to reduce the carry over effect, the PB-ARS questions during the lectures were not similar to the MCQs sheet. The used MCQs were piloted between authors to ensure its content validity and reliability. Contents validity was tested using test matrix and expert judgment. The test reliability was estimated using inter-rater reliability, a correlation of more than 0.7 was considered acceptable.

Summative exam:

Both groups attended their final written summative exams. L1 was undertaken 11 weeks prior to final exam while L2 was undertaken 10 weeks before the exam. The final exam was in MCQs format and included questions from all subjects taught in the second semester of the year including five questions relevant to the subjects taught in L1 and L2. The exam questions were identical for all students and were delivered at the same time under controlled conditions. Students who failed to attend the final summative exam were excluded to reduce the effect of time factor as confounding factors. The final exam scores of all student to questions related to TL1 and TL2 were anonymously collated using an excel sheet by independent tutor to reduce reporting bias. The maximum achievable score for the five questions relevant to the subjects taught in L1 and L2 was 5.

Students' perception:

At the end of L1, both groups were asked to fill a questionnaire regarding their experience with the lecture and intervention group participants were asked specific questions about their experience with PA-ARS . The used questionnaire was modified version from a previously used questionnaire to assess students experience with ARS in a recent trial . Students' responses were saved in an excel sheet after each lecture (L1, L2).

Analysis of the results:

Students' scores were saved in an excel sheet after each test. A specialized statistical analysis software was used (IBM SPSS statistics 22, version 22) The statistician was blinded to the allocation group. Scores were analyzed and compared to assess knowledge retention using cross-over analysis with Mann-Whitney U test for pre and post lecture quiz and t-test for summative test.

ELIGIBILITY:
Inclusion Criteria:

fourth-year undergraduate dental student

Exclusion Criteria:

Other undergraduate dental students from levels other than the 4th

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2018-05-29 (Actual)

PRIMARY OUTCOMES:
Formative exam | 10 minutes
  MCQs formative tests consisted of 20 questions related to the taught topics during L1 and L2 was undertaken

SECONDARY OUTCOMES:
Perception | 10 minutes
  At the end of L1, both groups were asked to fill a questionnaire regarding their experience with the lecture and intervention group participants were asked specific questions about their experience with PA-ARS

CONTACTS AND LOCATIONS:
Overall Officials: Fahad Alharbi, PhD, Principal Investigator — Prince Sattam Bin Abdulaziz University; Mohamed Almuzian, DClin.Dent.Orth, Study Chair — University of Edinburgh; Lubna Almuzian, DClin.Dent.Peado, Study Director — Berkeley Clinic at Glasgow
Locations (2):
- Saudi Arabia (2):
  - Prince Sattam Bin Abdulaziz University, Al Kharjah
  - Prince Sattam University, Riyadh

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR, Analytic Code
Time Frame: one year
Access Criteria: Any academic

REFERENCES:
- [Background] Dhaliwal HK, Allen M, Kang J, Bates C, Hodge T. The effect of using an audience response system on learning, motivation and information retention in the orthodontic teaching of undergraduate dental students: a cross-over trial. J Orthod. 2015 Jun;42(2):123-35. doi: 10.1179/1465313314Y.0000000129. Epub 2015 Apr 7. PMID 25849094